CLINICAL TRIAL: NCT00374465
Title: Prospective, Randomized Comparison of Therapy With Verapamil or Carvedilol on Long-Term Outcomes of Patients With Chronic Heart Failure Secondary to Non-Ischemic Cardiomyopathy
Brief Title: Therapy With Verapamil or Carvedilol in Chronic Heart Failure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Silesia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CavsBe.06
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: Dilated Cardiomyopathy
Keywords: Dilated Cardiomyopathy; Heart Failure
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure | interventions — Verapamil; Carvedilol

INTERVENTIONS:
Drug: Verapamil
Drug: Carvedilol

SUMMARY:
The aim of this study is to compare the effect of treatment with verapamil or carvedilol on long-term outcomes in stable, chronic heart failure secondary to non-ischemic cardiomyopathy.

DETAILED DESCRIPTION:
Heart failure, irrespective of its etiology may be viewed as a progressive disorder initiated by a different events and sustained by a multifaceted pathophysiological mechanisms. Regardless of the nature of the initiating events and optimized therapy used, loss of functioning cardiac myocytes developed and the disease progressed. One potential explanation for such progression is that not all pathological mechanisms underlying the disease are antagonized enough by currently used therapeutic strategy. Accordingly, impaired myocardial perfusion secondary to microvascular dysfunction has been postulated to play a major role in the progression of heart failure despite standard therapy for heart failure. It has been hypothesized that diffuse subendocardial ischemia due to altered coronary physiology may contribute to the global cardiac dysfunction seen in heart failure patients. Accordingly, coronary endothelial dysfunction at the microvascular and epicardial level in patients with acute-onset idiopathic dilated cardiomyopathy and chronic congestive heart failure has been reported. Thus, taking all mentioned above into account, the improvement in endothelial function and diminishing of subendocardial ischemia with calcium antagonists may be promising in terms of using these drugs for therapy of patients with stable chronic heart failure. The previous randomized study (5) and our long-term pilot study support this point of view.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure (NYHA II and III; LV ejection fraction, ≤ 35%) secondary to non-ischemic cardiomyopathy
* Stable condition at least 6 months before enrollment on conventional therapy (beta-blockers, ACE inhibitors and diuretics).

Exclusion Criteria:

* Improvement in clinical status on conventional therapy in out-patients period preceded hospitalization,
* Any changes narrowing epicardial coronary arteries in coronary angiography,
* Insulin dependent diabetes,
* Valvular heart disease (except the relative mitral regurgitation),
* Endocrine disease
* Significant renal and liver disease
* Alcohol abuse
* Lack of written informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-01; Study Completion 2008-05

PRIMARY OUTCOMES:
Sserum level of NT-proBNP,LVEF, LV diameters, exercise capacity (NYHA, V02,6 min walking test, changes in quality of life (MLHFQ).
In addition to secondary endpoints efficacy, patients will be classified as improved if they meet an increase of > 10 percentage points in the absolute EF and decrease in NT-proBNP levels at least 50% as compared with baseline study.

SECONDARY OUTCOMES:
Combined: mortality, heart transplantation, and readmission to hospital due to heart failure progression

CONTACTS AND LOCATIONS:
Overall Officials: Jan Wodniecki, Prof., Study Chair — Medical University of Silesia
Locations (1):
- Silesian Centre for Heart Disease, 3rd Department of Cardiology, Zabrze, Szpitalna 2 Saint, Poland